CLINICAL TRIAL: NCT00005736
Title: Interventions to Improve Asthma Management/Prevention at School
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4945
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
To design, develop, implement, and test the effectiveness of a three component health services and health education intervention for primarily Hispanic inner-city elementary school students at high risk for asthma morbidity and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of an initiative "Interventions to Improve Asthma Management and Prevention at School". The Broad Agency Announcement was released in June, 1994.

DESIGN NARRATIVE:

The study used a randomized intervention trial to test the effectiveness of a comprehensive school-based asthma program to increase linkages with primary care physicians, to increase self-management activities, and to reduce morbidity associated with asthma. The study used a nested design in which the schools were the unit of design, allocation, and analysis. Effects were measured from aggregate data about students and data from school measures to control asthma. There were three components to the intervention. First, case finding for asthma through screening in both intervention and control schools. Second, a linkage management system that connected the child with a source of primary care and enhanced communication among the school nurse, the primary care physician, and parents. Third, the development and implementation of interactive multimedia and decision support system techniques to tailor individualized learning opportunities for children with asthma. The interventions occurred in the school setting and included tailored feedback for children, teachers, nurses, primary care providers, and the family. Assessments were made of the potential for diffusion of the components to target audiences.

ELIGIBILITY:
Inclusion:

School-aged children enrolled at participating schools

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Guy Parcel — University of Texas

REFERENCES:
- [Background] Tortolero SR, Bartholomew LK, Tyrrell S, Abramson SL, Sockrider MM, Markham CM, Whitehead LW, Parcel GS. Environmental allergens and irritants in schools: a focus on asthma. J Sch Health. 2002 Jan;72(1):33-8. doi: 10.1111/j.1746-1561.2002.tb06509.x. PMID 11865797